CLINICAL TRIAL: NCT03416491
Title: Evaluation of Efficacy and Safety of KW-136 Plus Sofosbuvir for Treatment-naive Adults Chronically Infected With Hepatitis C Virus: a Randomized, Open-label, Multicenter Phase 2 Trial
Brief Title: Safety and Efficacy of KW-136 and Sofosbuvir for Treatment of Chronic Hepatitis C
Acronym: KW-136_II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kawin Technology Share-holding Co., Ltd. (Industry)
Collaborators: KawinGreen Biotech Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BJKY-2016-006; CTR20170073 (Registry Identifier: China Drug Trials)
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Hepatitis C, Chronic
Keywords: Chronic hepatitis C; Hepatitis C virus; KW-136; sofosbuvir; nonstructural protein 5A; nonstructural protein 5B; panogentypic regimen
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — Sofosbuvir

STUDY DESIGN:
Intervention Model Description: parallel, stratified assignment
Masking Description: The centralized laboratory was blinded to treatment assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NC_30 (Experimental): Non-cirrhotic subjects were medicated with KW-136 capsules 30 mg once daily and fixed-dose (400 mg once daily) sofosbuvir tablets for 12 successive weeks.
  Interventions: Drug: KW-136; Drug: Sofosbuvir
- NC_60 (Experimental): Non-cirrhotic subjects were medicated with KW-136 capsules 60 mg once daily and fixed-dose (400 mg once daily) sofosbuvir tablets for 12 successive weeks.
  Interventions: Drug: KW-136; Drug: Sofosbuvir
- LC_60 (Experimental): Cirrhotic subjects were medicated with KW-136 capsules 60 mg once daily and fixed-dose (400 mg once daily) sofosbuvir tablets for 12 successive weeks.
  Interventions: Drug: KW-136; Drug: Sofosbuvir

INTERVENTIONS:
Drug: KW-136 — KW-136 30 mg was provided in 3 capsules, 10 mg each, and KW-136 60 mg in a single capsule of 60 mg.
  Other Names: Coblopasvir
Drug: Sofosbuvir — Sofosbuvir was provided in a single tablet of 400 mg.

SUMMARY:
This study aimed to evaluate the safety and efficacy of KW-136, an investigational anti-hepatitis C virus (HCV) drug, combined with sofosbuvir for treatment of Chinese adults chronically infected with HCV. Thirty (30) non-cirrhotic subjects were medicated with KW-136 30 mg daily, 60 non-cirrhotic subjects with KW-136 60 mg daily, and 30 cirrhotic subjects with KW-136 60 mg daily; all the 120 subjects received sofosbuvir 400 mg daily. The treatment course lasted 12 successive weeks and thereafter all the study participants entered into a 12-week treatment-free follow-up period.

DETAILED DESCRIPTION:
It is estimated that China has a population of over 10 million infected with HCV and also a highly variable HCV genotype geographic distribution. A simple, universal, non-genotype-specific treatment regimen is preferred for anti-HCV treatment in clinical practice and public health. KW-136 and sofosbuvir are potent anti-HCV agents targeting at different HCV proteins, namely, nonstructural protein 5A and 5B, respectively. The combination regimen of KW-136 and sofosbuvir is expected to completely suppress HCV replication in subjects chronically infected with HCV and achieve a sustained virologic response, namely, HCV not detected or below a predefined limit in plasma, 12 or 24 weeks after cessation of treatment.

As KW-136 and sofosbuvir are both pan-genotypic anti-HCV agents (in simple words, effective for all known common genotypes of HCV), the combination of these two agents is also supposed to be efficacious for treatment of subjects chronically infected with HCV of all major genotypes and subtypes. An apparent clinical benefit of this pan-genotypic anti-HCV treatment regimen is that no complex, delicate HCV genotype sequencing is required before initiation of treatment to determine genotype-specific treatment alternatives of choice. This advantage is of great significance in the primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* aged between 18 and 65 years (inclusive) at the time of informed consenting and of either sex
* with a body mass index (BMI) between 18 and 30 kg/m^2 (inclusive)
* chronically infected with HCV, namely, with positive anti-HCV, HCV RNA or genotyping results at least six (6) months before the baseline, or with a liver biopsy confirming chronic hepatitis at most twelve (12) months before the baseline or during the screening period
* anti-HCV positivity and at least once testing result with HCV RNA equaling to or above 10^4 IU/mL
* genotyped to be gentoype (GT-1) or non-GT-1(including GT-2, 3, 6 or others) by the centralized laboratory
* naive to anti-HCV treatment, defined as being not previously treated with any interferon (including interferon alfa or beta or peginterferon), ribavirin, or other approved, investigational or any other not approved anti-HCV regimens of any source
* with or without cirrhosis (cirrhosis defined as FibroScan liver stiffness modulus (LSM) at least 14.6 kPa on screening, or liver biopsy confirming presence of cirrhosis within twelve (12) months before screening or within screening; no cirrhosis defined as FibroScan LSM below 14.6 kPa or liver biopsy confirming absence of cirrhosis within twelve (12) before screening or within screening; liver biopsy result takes priority over FibroScan LSM)
* women of childbearing potential (including postmenopausal women at or under 50 years of age) with negative blood pregnancy test results; subjects of childbearing potential (including male subjects and their female partners) have no childbearing plan from screening, initiation of treatment until six (6) months after end of treatment and consent to use effective contraceptive measures
* voluntary participation in the study and being able to understand and sign the informed consent form

Exclusion Criteria:

* having previously used any investigational or experimental direct antiviral agents against HCV, including protease, NS5B polymerase or NS5A inhibitors, before screening
* having received any interferon-based anti-HCV regimens before screening
* having been exposed to any systemic potent immunomodulators , such as steroids or thymosin alfa (excluding use of nasal, inhalational, topical steroids and/or others) for more than two weeks within six (6) months before screening, or anticipated to be exposed to these agents during the study period
* with hepatitis B virus surface antigen (HBsAg) or anti-human immunodeficient virus (HIV) positivity
* with evidence of decompensatory liver function, including but not limited to total serum bilirubin (TBIL) above twice (2) of the upper limit of normal (ULN), serum albumin (ALB) below 35 g/L, or prothrombin activity (PTA) below 60% confirmed on repeated testing; emergence of ascites, upper gastrointestinal bleeding and/or hepatic encephalopathy; with liver function reserve Child-Pugh class B or C
* with primary liver cancer confirmed or evidenced by serum alfa-fetoprotein above 100 ng/ml or liver imaging study showing suspected nodules
* with a previous history of liver disease of other causes, including alcoholic liver disease, nonalcoholic steatohepatitis, drug-induced hepatitis, autoimmune hepatitis, Wilson disease or hemochromatosis
* with serum alaine aminotransferase (ALT) or asparate aminotransferase (AST) above ten (10) times of ULN confirmed on repeated testing
* with white blood cell (WBC) count below 3x10^9 per liter, neutrophil count below 1.5x10^9 per liter (or below 1.25x10^9 per liter for cirrhotics), platelet count below 50x10^9 per liter, or hemoglobin below 120 g/L (for males) or 110 g/L (for females) confirmed on repeated testing
* with serum creatinine clearance (CLcr) below 50 ml/min using the Cockcroft-Gault formula confirmed on repeated testing
* with uncontrolled diabetes mellitus (hemoglobin A1c[HbA1c] above 7.0% confirmed on repeated testing)
* with psychiatric or neurologic disorders, including previous or family history of psychiatric disorders (especially depression, depressive state, epilepsy or hysteria)
* with serious cardiovascular disorders, including uncontrolled hypertension (systolic blood pressure at or above 160 mmHg and/or diastolic blood pressure at or above 100 mmHg), heart insufficiency of New York Heart Association class III or above, history of myocardial infarction within six (6) months before screening, history of percutaneous transluminal coronary angioplasty within six (6) months before screening, unstable angina pectoris, QTc interval (Fridericia correction formula QTc = QTxRR^-1/3) at or above 450 msec or second- or third-grade atrioventricular block or any other uncontrolled arrhythmias confirmed on repeated electrocardiography on screening
* with serious hematologic disorders (such as anemia, hemophilia and others)
* with serious kidney diseases (such as chronic kidney disease, kidney insufficiency and others)
* with serious gastrointestinal disorders (such as peptic ulcer, colitis and others)
* with serious respirator disorders (such as active pulmonary tuberculosis, lung infection, chronic obstructive pulmonary disease, pulmonary interstitial disease and others)
* with active or suspected malignant tumors or with a previous history of malignant tumors (excluding skin basal cell carcinoma or cervical carcinoma in situ) within five (5) years before screening
* with a history of major organ transplantation
* being known to be severely hypersensitive or allergic to any drugs, especially the testing medications and other constituents
* with a history of active alcohol or drug abuse within six (6) months before screening
* being pregnant or lactating
* being unable to discontinue prohibited medications as defined by the protocol
* having participated in any other clinical studies within three (3) months before screening
* being unable or unwilling to provide informed consent or unable to follow the protocol requirements
* any other conditions of excluding a potential participant at the discretion of the investigators

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-09-17 (Actual); Study Completion 2017-11-08 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response at 12 weeks after end of treatment (SVR12) | 12 weeks after end of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)

SECONDARY OUTCOMES:
Sustained virologic response at 4 weeks after end of treatment (SVR4) | 4 weeks after end of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 1 week after initiation of treatment (RVR1) | 1 week after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 2 weeks after initiation of treatment (RVR2) | 2 weeks after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 4 weeks after initiation of treatment (RVR4) | 4 weeks after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 8 weeks after initiation of treatment (RVR8) | 8 weeks after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)
Rapid virologic response at 12 weeks after initiation of treatment (RVR12) | 12 weeks after initiation of treatment
  Percentage of subjects with plasma HCV not detected or below the lower limit of quantitation (15 IU/mL)

OTHER OUTCOMES:
Virologic breakthrough | 2, 4, 8 and 12 weeks after initiation of treatment
  Percentage of subjects with on-treatment re-detected plasma HCV RNA after HCV RNA below the lower limit of quantitation
Virologic relapse | 4 and 12 weeks after end of treatment
  Percentage of subjects with off-treatment re-detected plasma HCV RNA after end-of-treatment HCV RNA below the lower limit of quantitation

CONTACTS AND LOCATIONS:
Overall Officials: Lai Wei, M.D., Principal Investigator — Peking University People's Hospital
Locations (12):
- China (12):
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - Capital Medical University Affiliated Beijing Youyi Hospital, Beijing, Beijing Municipality
  - Capital Medical University Affiliated Beijing You'an Hospital, Beijing, Beijing Municipality
  - Chinese PLA Third Military Medical University First Affiliated Hospital, Chongqing, Chongqing Municipality
  - Guangzhou Municipal Eighth People's Hospital, Guanzhou, Guangdong
  - He'nan Provincial Hospital of Infectious Disease (Zhengzhou Municipal Sixth People's Hospital), Zhengzhou, He'nan
  - Nanjing Municipal Second Hospital, Nanjing, Jiangsu
  - Jilin University First Hospital, Changchun, Jilin
  - Dalian Municipal Sixth People's Hospital, Dalian, Liaoning
  - Shenyang Municipal Sixth People's Hospital, Shenyang, Liaoning
  - Ji'nan Municipal Hospital of Infectious Disease, Ji'nan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong

IPD SHARING:
Plan to Share IPD: No
No IPD plan is included in the study protocol.

REFERENCES:
- [Derived] Rao H, Song G, Li G, Yang Y, Wu X, Guan Y, Mao Q, Jiang X, Wang C, Zhang Y, Jia J, Guo X, Li C, Ning J, Qin H, Pan H, Wei L. Safety and efficacy of coblopasvir and sofosbuvir in patients with genotypes 1, 2, 3 and 6 HCV infections without or with compensated cirrhosis. J Viral Hepat. 2020 Jan;27(1):45-51. doi: 10.1111/jvh.13208. Epub 2019 Oct 2. PMID 31520460